CLINICAL TRIAL: NCT06291766
Title: The Impact of Continous Glucose Monitoring on Pregnancy Outcome, in Women With Gestational Diabetes and a History of Gastric Bypass Surgery.
Brief Title: Gestational Diabetes After Gastric Bypass Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Ulrika Moll, MD, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-05498-01
Record Dates: First submitted 2024-02-05; First posted 2024-03-04 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-02

CONDITIONS: Diabetes, Gestational; Gastric Bypass Status for Obesity Complicating Pregnancy, Childbirth, or the Puerperium; Pregnancy in Diabetic; Blood Glucose Self Monitoring
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continous glucose measurement (Other): Use of FreeStyle Libre 3, with Libre Link app and Glooko app for measurement and review of glucose measurements.
  Interventions: Device: FreeStyle Libre 2, continous glucose monitoring
- Capillary glucose measurement (No Intervention): Standard care, including capillary glucose measurements and Glooko app for review of glucose measurements.

INTERVENTIONS:
Device: FreeStyle Libre 2, continous glucose monitoring — The use of FreeStyle Libre 3 sensors and Libre Link app and Glooko app for analysing glucose control in pregnancy
  Arms: Continous glucose measurement

SUMMARY:
The goal of this trial is to compare different means of glucose monitoring in women with gestational diabetes and a history of gastric bypass surgery.

The main question it aims to answer is:

How does continous glucose monitoring impact the treatment and affect pregnancy outcome in these women.

Participants will be randomized to either continous glucose monitoring or regular capillary glucose measurements during the last trimester of their pregnancy. Researchers will compare the glucose measurement outcomes, the glucose lowering treatment given and pregnancy outcomes between groups.

DETAILED DESCRIPTION:
The project aims to investigate gestational diabetes in women with a history of gastric bypass surgery (GBP). The investigators will analyse glucose levels by using continuous glucose measurement (GCM) or capillary glucose measurements and compare mean glucose values, treatment and the pregnancy outcome.

In Sweden the incidence of gestational diabetes is 2-5% of pregnancies, but the frequency varies greatly in different areas and in different ethnicities. The women with gestational diabetes have an increased risk of complications during pregnancy. The most acknowledged complications are large for gestational age infants (LGA), preeclampsia and caesarean section. The infants have a higher need for neonatal intensive care, due to the risk of hypoglycaemia, hypoxia and jaundice postpartum. Treating gestational diabetes and normalizing glucose values have been proven to reduce risks of unfavourable pregnancy outcome.

Gastric bypass surgery is a common treatment for obesity. The frequency of young women with gastric bypass surgery and concomitant gestational diabetes have increased. Many maternity care centres have started to use a 3-7 day screening for gestational diabetes, since the routine oral glucose toleration test (OGTT) is not recommended after GBP. It is previously shown that women with GBP have a decreased risk of GDM and LGA infants. However, there is an increased risk of small for gestational age (SGA). There is a lack of knowledge and guidelines regarding the optimal treatment of gestational diabetes in these women. How the glucose variability affects pregnancy outcome is poorly investigated. At Lund University Hospital, Region Skane, Sweden, the screening procedure used since 2012 for GDM-screening in women with GBP is a 3 day 7-point capillary glucose measurement. Approximately 25% of the pregnant women with GBP is diagnosed with GDM, using this method at Lund University Hospital.

In this project the investigators will randomize women with gestational diabetes and a history of gastric bypass (GDM-GBP) into two different groups in the last trimester of pregnancy. Both groups are given standard medical care, which includes visits to the Specialized Maternity Care Unit and weekly follow up by the diabetologist. The first group is given continuous glucose measurement (FreeStyle Libre3) and the other group is given standard medical care which includes 7-point capillary glucose measurement. With the CGM system it is possible to collect more comprehensive data regarding glucose values and variability. Previous studies have shown that women with gastric bypass surgery have an earlier than normal postprandial glucose excursion and are more prone to later postprandial hypoglycaemia. During this study, the physician as well as the patient can observe the early glucose excursion after meals and measure time in target, time above target and time below target. Large for gestational age and accelerated growth of the infant is supposed to be due to high glucose values and a high proportion of Time above target. The increased risk of SGA infants in these women is hypothesized to be due to a large proportion of time below target. However, this theory is not sufficiently investigated and it is not known if the use of CGM can help to reduce the risk of weight deviation in the infants.

The investigators want to examine if new technique in glucose measurement can contribute to more favourable pregnancy outcome in women with gestational diabetes and a history of GDM. The main question is if the use of CGM affect pregnancy outcome. The secondary outcomes includes glucose variability and the use of different treatment approaches in GDM in this group of women.

ELIGIBILITY:
Inclusion Criteria:

* Understands written and spoken Swedish
* Previous Gastric Bypass surgery
* Diagnosed with gestational diabetes according to our local criteria
* Planned follow up at the Specialized Maternity Ward at Skane University Hospital
* Understands the use of CGM and is willing to use the system
* Have signed informed consent

Exclusion Criteria:

* Other kinds of bariatric surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Pregnancy Outcome | During delivery and postpartum (measured up to 5 days postpartum)
  ANY: Caesarian section (Y/N), instrumental delivery (Y/N), preeclampsia (Y/N), premature birth before week 37 (Y/N), Macrosomia (>4000g) (Y/N), Large for gestational age infant (Y/N), small for gestational age infant (Y/N), shoulder dystocia (Y/N), neonatal hypoglycemia (Y/N) (<4 hours after birth: <1.4 mmol/L; 4 to <24 hours after birth: <1.9 mmol/L; 24 to <48 hours after birth: <2.8 mmol/L, ≥48 hours after birth: 3.3 mmol/L

SECONDARY OUTCOMES:
Glucose values | Gestational week 28-42
  Mean/median glucose values (mmol/l)
Glucose values | Gestational week 28-42
  Glucose variability (SD)
Glucose values | Gestational week 28-42
  % Time in Target (3,5-7,8 mmol/l)
Glucose values | Gestational week 28-42
  % Time below target
Glucose values | Gestational week 28-42
  % Time above target
Pharmacological treatment | Gestational week 28-42
  The use of insulin (Y/N)
Pharmacological treatment | Gestational week 28-42
  the dose of insulin (IE)
Pharmacological treatment | Gestational week 28-42
  the use of Metformin (Y/N)
Pharmacological treatment | Gestational week 28-42
  the dose of metformin (g/day)
Birthweight | at the day of birth
  birth weight of infant (g)
Week of delivery | exact day (ie 28+0 to 42+6)
  gestational week

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Moll, MD, PhD, Principal Investigator — Region Skane
Locations (1):
- Region Skane, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moll U, Landin-Olsson M, Nilsson C, Ursing D, Strevens H. Pregnancy outcome in women with gestational diabetes - A longitudinal study of changes in demography and treatment modalities. Acta Obstet Gynecol Scand. 2020 Mar;99(3):333-340. doi: 10.1111/aogs.13758. Epub 2019 Dec 22. PMID 31654523